CLINICAL TRIAL: NCT02102828
Title: Efficacy of Prolonged Distal Calf Compression as Part of a Multimodal DVT Protocol in Tourniquet-less Total Knee Arthroplasty: a Randomized Clinical Trial in 100 Patients
Brief Title: Multimodal DVT Protocol in Tourniquet-less Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14045-14-008
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2015-10

CONDITIONS: Deep Vein Thrombosis
Keywords: DVT; Total Knee Arthroplasty
MeSH Terms: conditions — Venous Thrombosis | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin only (Placebo Comparator): Patients receive aspirin therapy
  Interventions: Other: Aspirin
- extended compression (Experimental): aspirin and extended compression therapy in combination
  Interventions: Device: extended compression

INTERVENTIONS:
Device: extended compression — Home use of extended compression therapy and aspirin
  Arms: extended compression
Other: Aspirin — standard therapy of aspirin
  Arms: Aspirin only

SUMMARY:
The Cothera VPulse(tm) mechanical compression device (MCD) combines rapid intermittent sequential compression with cold therapy and is designed for single patient use in the home. Additionally, it can track patient compliance. This study will examine if there is a difference in deep vein thrombosis (DVT) occurrence over 3 weeks after tourniquet-less total knee arthroplasty (TKA) and multimodal prophylaxis with or without extended MCD use in a cooling device/MCD system.

DETAILED DESCRIPTION:
In recent years there has been significant progress towards more effective and practical thromboprophylaxis in joint replacement surgeries. Since Aspirin 325mg twice daily has been recently included as a nationally approved venous thromboembolism (VTE) prophylaxis in the Surgical Care Improvement Project (SCIP) protocols for low risk total knee arthroplasty (TKA) patients, it is necessary to optimize multimodal prophylaxis methods. These include reduced tourniquet time, early mobilization, and mechanical compression devices (MCDs). MCDs are commonly used as part of the in-hospital VTE prophylaxis measures; however, it has not been demonstrated in clinical trials that optimal prophylaxis methods would be enhanced by prolonged use of a MCD after discharge. In order to achieve this, a potentially valuable solution has recently been made available to the outpatient population. The Cothera VPulse(tm) is a MCD that combines rapid intermittent sequential compression with cold therapy. It is designed for single patient use in the home and includes technology to track patient compliance. The purpose of this study is to examine if there is a difference in DVT occurrence over 3 weeks after tourniquet-less TKA and multimodal prophylaxis with or without extended MCD use in a cooling device/MCD system.

ELIGIBILITY:
Inclusion Criteria:

* TKA candidacy, osteoarthritis, patients able to understand study intent, and agree to study participation

Exclusion Criteria:

* Subjects with personal or family history of DVT, currently taking antiplatelet/anticoagulant drugs, genetic risk factor positive for VTE, pronounced thrombocytopenia, GI bleed within 6 months of surgery, NSAID intolerance, orthopaedic and medical co-morbidities that would prevent postoperative rapid mobilization and compliance with MCD such as extra-articular pathology with referred pain to the knee (spinal stenosis, neuropathy, ipsilateral hip disease), severe knee deformity, post-traumatic and inflammatory arthritis, BMI above 40, active knee sepsis, remote sites of active infection, ASA class > lll, cardiac disease failing medical clearance, severe liver disease, peripheral artery disease, seizure disorder, alcohol abuse, smoking abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
DVT Occurence | 3 weeks
  DVT Occurence measured by physical assessment and duplex ultrasound images for DVT detection

SECONDARY OUTCOMES:
Patient Satisfaction | 10 days
  Patient satisfaction will be measured 10 days postop using the EuroQol standardized instrument
Mobilization | 10 days
  Patient activity level will be measured using the standardized UCLA Activity Score

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Snyder, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- Good Samaritan Hosptial, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Snyder MA, Sympson AN, Scheuerman CM, Gregg JL, Hussain LR. Efficacy in Deep Vein Thrombosis Prevention With Extended Mechanical Compression Device Therapy and Prophylactic Aspirin Following Total Knee Arthroplasty: A Randomized Control Trial. J Arthroplasty. 2017 May;32(5):1478-1482. doi: 10.1016/j.arth.2016.12.027. Epub 2016 Dec 23. PMID 28159420